CLINICAL TRIAL: NCT02302235
Title: Ketogenic Diet Treatment Adjunctive to Radiation and Chemotherapy in Glioblastoma Multiforme: a Pilot Study
Acronym: GBMXRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Collaborators: Neuroscience Research Foundation, Sewickley,PA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: maesc 006
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: Glioblastoma multigorme; Ketogenic Diet; radiotherapy; chemotherapy; safety; efficiency
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketogenic Diet (Active Comparator): Treatment will consist of ketogenic diet. KGD will consist of 4:1 [fat] : [protein+carbohydrate] weight ratio with 1600 kcal restriction. Diet will be started at the time of initiation of radiation treatment.
  Interventions: Other: Standardized Diet
- Standardized diet (Other): The subjects will be taken standard diet in a 1:1 ratio.
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — Treatment will consist of ketogenic diet. KD will consist of 4:1 [fat] : [protein+carbohydrate] weight ratio with 1600 kcal restriction.
  Other Names: KGD
  Arms: Standardized diet
Other: Standardized Diet — Participants with GBM treated with radiation and temozolomide after surgical debulking treatment. The subjects will be taken standard diet in a 1:1 ratio. Diet will be started at the time of initiation of radiation treatment.
  Arms: Ketogenic Diet

SUMMARY:
The goal of the present study is to evaluate efficacy, safety and tolerability of 4:1 ketogenic diet administered adjunctively to standard radiation and temozolomide chemotherapy in patients with GBM in a prospective, randomized open label study.

DETAILED DESCRIPTION:
Primary aims of the study will be to 1) To evaluate efficacy of ketogenic diet as adjunctive treatment of radiation treatment in glioblastoma multiforme. 2) To evaluate the safety of ketogenic diet as adjunctive treatment of radiation treatment in glioblastoma multiforme. Secondary aim will be to evaluate tolerability of ketogenic diet as adjunctive treatment of radiation treatment in glioblastoma multiforme.

Participants will be seen at one, 2 weeks, and 4 weeks after KG diet initiation, and then monthly until month 6 after diet initiation, then every 2 months until 2 years after treatment initiation or death, then every 3 months until 3 years after treatment initiation or death. KD treatment will last for 6 months or until exit criteria are met, whichever comes first. Exit criteria are the primary outcome measures, the first of either (a) MRI tumor progression or (b) death. Secondary outcome measures will include treatment compliance, hunger scale scores, fasting serum glucose and BOH levels and occurrence of adverse events.

Patients with documented tumor progression will receive standard care for progressive GBM as directed by their treating oncologist, independent of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Ability and willingness to signed informed consent form
3. Astrocytoma grade 4 (glioblastoma multiforme, GBM, histologically confirmed, WHO criteria)
4. Documented surgical resection/debulking
5. Measurable contrast-enhancing GBM by MRI imaging ≤ two weeks before screening or prior to surgery if done ≤ 2 months before
6. Karnovsky Performance Score of 70 or more

Exclusion Criteria:

1. Acute intracranial or intratumoral hemorrhage > Grade 1 either by MRI or CT scan ≤2 weeks of screening. (Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin may enter the study)
2. Prior treatment with any of the following: (a) small-molecule kinase inhibitor; (b) non-cytotoxic hormonal agent; (c) KD ≤6 months of enrollment
3. Planned continued use of glucocorticoids
4. Anticoagulation treatment with ≥ 1 mg/day coumadin ≤ 7 days prior to screening (low-dose [≤ 1 mg/day] coumadin, heparin, and low-molecular-weight heparin are permitted)
5. Any systemic illness or unstable medical condition that might pose additional risk, including: cardiac, unstable metabolic or endocrine disturbances, renal or liver disease, past history of renal calculi, hyperuricemia, hypercalcemia, mitochondrial disease, known disorder of fatty acid metabolism, porphyria, carnitine deficiency and pancreatitis
6. History of non-glioma malignancy other than:

   1. Surgically excised non-melanoma skin cancer or in situ carcinoma of the cervix
   2. A malignancy diagnosed ≥2 years ago if the subject has had no evidence of disease for 2 years prior to screening
7. History of uncontrolled hyperlipidemia
8. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements
9. History of human immunodeficiency virus, or hepatitis C
10. Failure to recover from <CTCAE grade 2 toxicities related to prior therapy
11. Pregnancy or breastfeeding
12. Use of any investigational drug within 1 months of enrollment
13. Inability or unwillingness of subject to give written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-02; Primary Completion 2021-12 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
survival time | 6 months
  We hope to achieve a substantial difference in both survival time and time to recurrence between the KD and non-KD treatment groups. Survival time of 3 years from treatment initiation and tumor progression-free time of 2.5 years from treatment initiation would be extraordinary compared to historical data.
time to radiological (MRI) tumor progression | 6 months
  MRI outcome will be assessed by the radiographic assessment in neuro-oncology criteria based on contrast-enhanced cranial MRI scans evaluating measureable disease, measured as the sum of products of perpendicular diameters (bi-dimensional measurements) of all measurable enhancing lesions and non-measurable disease.
The incidence of treatment-emergent adverse events during treatment | 6 months
  Incidence of treatment-emergent adverse events changes in laboratory evaluations, changes in physical examination findings will be compared between the KD and control treatment groups

SECONDARY OUTCOMES:
Tolerability of ketogenic diet: Rate of early discontinuation of subjects from the diet because of intolerability, defined as unwillingness by the subject to continue with the diet because of possible diet related side effects | 6 months
  Rate of early discontinuation of subjects from the diet because of intolerability, defined as unwillingness by the subject to continue with the diet because of possible diet related side effects will be evaluated using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, M.D., Principal Investigator — Mid-Atlantic Epilepsy and Sleep Center
Locations (1):
- MidAtlantic Epilepsy and Sleep Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Klein P, Tyrlikova I, Zuccoli G, Tyrlik A, Maroon JC. Treatment of glioblastoma multiforme with "classic" 4:1 ketogenic diet total meal replacement. Cancer Metab. 2020 Nov 9;8(1):24. doi: 10.1186/s40170-020-00230-9. PMID 33292598